CLINICAL TRIAL: NCT04746183
Title: AGILE: Seamless Phase I/IIa Platform for the Rapid Evaluation of Candidates for COVID-19 Treatment
Brief Title: AGILE (Early Phase Platform Trial for COVID-19)
Acronym: AGILE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); Royal Liverpool University Hospital (Other Government); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UoL001542i, UoL001542j
Record Dates: First submitted 2020-10-13; First posted 2021-02-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Covid19
Keywords: SARS coronavirus 2; SARS-CoV-2; Phase I; Phase II; Platform trial
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir; nitazoxanide; VIR-7832; sotrovimab; favipiravir; nirmatrelvir and ritonavir drug combination; remdesivir; Ritonavir

STUDY DESIGN:
Intervention Model Description: CST2: Closed CST3A: Closed CST3B: Closed CST5: Closed CST6: Closed CST8: Closed CST9a:1:1:1 randomised open label Phase II of ALG-097558 versus ALG-097558+ remdesivir VS SOC CST9b: Double Blind 1:1 stratified randomised controlled adaptive trial with twice daily (Q12H) oral dose of ALG-097558 versus matching placebo for ALG097558.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: CST-2: Phase I, open-label EIDD-2801 vs standard of care. Phase II, blinded controlled parallel group of EIDD-2801 vs placebo CST-3A: Phase Ia, open-label nitazoxanide CST-3B: Phase Ib, II, open label nitazoxanide vs standard of care CST-5: Phase I, blinded VIR-7832 vs placebo, Phase II, blinded VIR-7832 vs VIR-7831 vs placebo CST-6: Open label IV favipiravir vs standard of care CST-8: Open label Molnupiravir and Paxlovid® versus standard of care CST-9a: Open label ALG-097558 versus ALG-097558 + remdesivir versus standard of care CST-9b:Double Blind ALG-097558 versus matching placebo for ALG097558
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (21):
- CST-2 EIDD-2801 Phase Ib (Experimental): EIDD-2801 (also known as MK-4482, molnupiravir). Phase Ib: EIDD-2801 will be administered orally, twice daily (BID) for 10 doses (5 or 6 days). The starting dose will be established based on safety and pharmacokinetics from the EIDD-2801-1001-US/UK study, and dose escalations may occur as described in this CST.
  Interventions: Drug: CST-2: EIDD-2801
- CST-2 Control (No Intervention): Phase 1b only (standard of care)
- CST-2 Placebo (Placebo Comparator): Phase II placebo blinded controlled
  Interventions: Drug: CST-2: Placebo
- CST-3A Nitazoxanide (Experimental): Phase Ia Nitazoxanide will be administered orally, initially twice daily (BID) for 14 doses (7 days). The starting dose will be 1500mg BID based on existing dose information, but dose adaptations may occur
  Interventions: Drug: Nitazoxanide
- CST-5 VIR-7832 Phase I (Experimental): Phase I: Single doses of VIR-7832 will be administered by intravenous (IV) infusion. The starting dose will be 50 mg, and dose escalations of 150 and 500 mg are anticipated.
  Interventions: Drug: VIR-7832
- CST-5 VIR-7831 Phase II (Active Comparator): Phase II: 500 mg dose of VIR-7831 will be given by IV infusion.
  Interventions: Drug: VIR-7831
- CST-5 Placebo Phase I (Placebo Comparator): Phase I: placebo blinded controlled
  Interventions: Drug: CST-5: Placebo
- CST3B Nitazoxanide (Experimental): Phase II experimental arm.
  Interventions: Drug: Nitazoxanide
- CST3B Control (No Intervention): Standard of care
- CST6 IV Favipiravir (Experimental): IV Favipiravir twice daily for 7 days. Starting dose 600 mg twice daily. Dose escalation to 1200 mg twice daily, 1800 twice daily, 2400 twice daily.
  Interventions: Drug: Favipiravir
- CST6 Control (No Intervention): Standard of care
- CST-2 EIDD-2801 Phase II (Experimental): EIDD-2801 (also known as MK-4482, molnupiravir).
  Phase II: As per Phase Ib, with the dose determined by the recommended phase II dose.
  Interventions: Drug: CST-2: EIDD-2801
- CST-8 Phase I Molnupiravir + Paxlovid® (Experimental): Molnupiravir 800mg Twice a day (BD) in combination with Paxlovid® (300mg nirmatrelvir + ritonavir 100mg) twice a day (BD) for 5 days as starting dose, with a de-escalation protocol reducing in increments of molnupiravir to 600mg BD, then 400mg BD if required. The dose of Paxlovid® will be fixed for all cohorts.
  Interventions: Drug: Molnupiravir; Drug: Paxlovid
- CST-8 Phase I Molnupiravir + Paxlovid® Control (No Intervention): Standard of care
- CST-5 VIR-7832 (Active Comparator): Phase II: 500 mg dose of VIR-7832 will be given by IV infusion.
  Interventions: Drug: VIR-7832
- CST-5 Placebo Phase II (Placebo Comparator): Phase II: placebo blinded controlled
  Interventions: Drug: CST-5: Placebo
- CST-9a Monotherapy (Experimental): Phase II: ALG-097558 600 mg twice a day orally for 5 days
  Interventions: Drug: ALG-097558
- CST-9a Combination (Experimental): Phase II: ALG-097558 600 mg twice a day orally for 5 days in combination with IV remdesivir for 3 days (200 mg day 1, 100 mg day 2 and 3)
  Interventions: Drug: ALG-097558; Drug: ALG-097558 and Remdesivir
- CST-9a Control (Active Comparator): Phase II : standard of care
  Interventions: Drug: NHS standard of care as per COVID-19 treatment guidelines
- CST-9b: ALG-097558 (Experimental): twice daily dose for 5 days
  Interventions: Drug: ALG-097558
- CST-9b: placebo for ALG097558 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CST-2: EIDD-2801 — CST-2 Phase Ib: EIDD-2801 will be administered orally, twice daily (BID) for 10 doses (5 or 6 days). The starting dose will be established based on safety and pharmacokinetics from the EIDD-2801-1001-US/UK study, and dose escalations may occur as described in this CST.
  Phase II: As per Phase Ib, with the dose determined by the recommended phase II dose.
  Other Names: MK-4482; Molnupiravir
  Arms: CST-2 EIDD-2801 Phase II; CST-2 EIDD-2801 Phase Ib
Drug: CST-2: Placebo — CST-2 Phase II: Placebo will be administered orally, twice daily (BID) for 10 doses (5 or 6 days).
  Other Names: Placebo
  Arms: CST-2 Placebo
Drug: Nitazoxanide — CST3A & CST3B Phase I: Nitazoxanide will be administered orally, initially twice daily (BID) for 14 doses (7 days). The starting dose will be 1500mg BID based on existing dose information, but dose adaptations may occur.
  Phase II: As per Phase Ib, with the dose determined by the recommended phase II dose.
  Arms: CST-3A Nitazoxanide; CST3B Nitazoxanide
Drug: VIR-7832 — CST-5: Phase I, Single doses of VIR-7832 will be administered by intravenous (IV) infusion over 1 hour. The starting dose will be 50 mg, and dose escalations of 150 and 500 mg are anticipated, with escalation guided by emerging safety data and decision by the SRC.
  Phase II: As per Phase I, with the dose determined by the recommended phase II dose.
  Arms: CST-5 VIR-7832; CST-5 VIR-7832 Phase I
Drug: VIR-7831 — CST-5 Phase II: A 500 mg dose of VIR-7831 will also be given by IV infusion over 1 hour.
  Other Names: Sotrovimab
  Arms: CST-5 VIR-7831 Phase II
Drug: CST-5: Placebo — CST-5 Phase 1, Phase II: Placebo given by intravenous infusion over 1 hour
  Other Names: Placebo
  Arms: CST-5 Placebo Phase I; CST-5 Placebo Phase II
Drug: Favipiravir — CST-6: Multiple doses of IV Favipiravir will be administered by intravenous (IV) infusion over 1 hour. Dosing regimen will be every 12 hours for 7 days duration. The starting dose will be 600mg (BID), and dose escalations to 1200mg (BID), 1800mg (BID) and 2400mg (BID) are anticipated as well as a de-escalation dose of 300mg (BID) if necessary, with de-escalation and escalation guided by emerging safety data and decision by the Safety Review Committee (SRC).
  Arms: CST6 IV Favipiravir
Drug: Molnupiravir — Molnupiravir 800mg Twice a day (BD) for 5 days as starting dose, with a de-escalation protocol reducing in increments of molnupiravir to 600mg BD, then 400mg BD if required.
  Other Names: Lagevrio
  Arms: CST-8 Phase I Molnupiravir + Paxlovid®
Drug: Paxlovid — Paxlovid® (300mg nirmatrelvir + ritonavir 100mg) twice a day (BD) for 5 days. The dose of Paxlovid® will be fixed for all cohorts.
  Other Names: nirmatrelvir and ritonavir
  Arms: CST-8 Phase I Molnupiravir + Paxlovid®
Drug: ALG-097558 — ALG-097558 600 mg Twice a day (BD) for 5 days
  Arms: CST-9a Combination; CST-9a Monotherapy
Drug: ALG-097558 and Remdesivir — ALG-097558 600 mg Twice a day (BD) for 5 days Remdesivir will be administered once daily by intravenous infusion over 30 to 120 minutes. 200 mg will be given on day 1 and 100 mg on day 2 and day 3.
  Other Names: ALG-097558 and veklury
  Arms: CST-9a Combination
Drug: NHS standard of care as per COVID-19 treatment guidelines — NHS standard of care as per COVID-19 treatment guidelines
  Other Names: any of the following: nirmatrelvir plus ritonavir (Paxlovid) sotrovimab (Xevudy) molnupiravir (Lagevrio)
  Arms: CST-9a Control
Drug: ALG-097558 — twice daily (Q12H) oral dose of ALG-097558
  Arms: CST-9b: ALG-097558
Drug: Placebo — twice daily (Q12H) oral dose
  Arms: CST-9b: placebo for ALG097558

SUMMARY:
The AGILE platform master protocol allows incorporation of a range of identified and yet-to-be-identified candidates as potential treatments for adults with COVID-19 into the trial. Candidates will be added into the trial via candidate-specific trial (CST) protocols of this master protocol as appendices. Having one master protocol ensures different candidates are evaluated in the same consistent manor and opening up new trials for new candidates is more efficient. Inclusion of new candidates will be based on pre-clinical data, evidence in the clinical setting and GMP capabilities.

DETAILED DESCRIPTION:
AGILE is a multicentre, multi-arm, multi-dose, multi-stage open-label, adaptive, seamless phase I/II Bayesian randomised platform trial to determine the optimal dose, activity and safety of multiple candidate agents for the treatment of COVID-19.

This study allows for the assessment of many candidates at different doses, with the ability to add candidates as they are identified or drop them as their evaluation is completed. Promising candidates will move to an external trial for further evaluation in the phase II/III setting.

Each candidate will be evaluated in its own trial, randomising between candidate and control with 2:1 allocation in favour of the candidate. Each dose will be assessed for safety sequentially in cohorts of 6 patients. Once a phase II dose has been identified we will assess efficacy by seamlessly expanding into a larger cohort.

AGILE is completely flexible in that the core design in the master protocol (as has been explained above) can be adapted for each candidate based on prior knowledge of the candidate - i.e. population, primary endpoint and sample size can be amended. This will be detailed in each candidate-specific trial protocol of the master protocol.

Candidate-Specific Trial 2 (CST-2): Open-label 2:1 randomised controlled phase I of EIDD-2801 versus standard of care followed by a 1:1 blinded controlled parallel group Phase II trial of EIDD-2801 versus placebo. A phase I will be carried out to confirm the optimal dose in this group. Following a safety review, EIDD-2801 will be tested for efficacy in a blinded placebo controlled randomised phase II trial.

Candidate-Specific Trial 3 (CST-3A): Multicentre, Adaptive, Phase I trial to Determine the optimal dose, Safety and Efficacy of Nitazoxanide for the Treatment of COVID-19

Candidate-Specific Trial 3 (CST-3B): A Randomized, Multicentre, Seamless, Adaptive, Phase I/II trial to Determine the optimal dose, Safety and Efficacy of Nitazoxanide for the Treatment of COVID-19

Candidate-Specific Trial 5 (CST-5): Randomized, Multicentre, Seamless, Adaptive, Phase I/II Platform Study to Determine the Phase II dose of VIR-7832, and Evaluate the Safety and Efficacy of VIR-7831 and VIR-7832 for the Treatment of COVID-19

Candidate-Specific Trial 6 (CST-6): A Randomized, Multicentre, Seamless, Adaptive, Phase I/II Platform Study to Determine the Phase II dose and to Evaluate the Safety and Efficacy of intravenous Favipiravir for the Treatment of COVID-19

Candidate-Specific Trial 8 (CST-8): A Randomised, Multicentre, Seamless, Adaptive, Phase I Platform Study to Determine the recommended Phase II dose and Evaluate the Safety and Efficacy of antiviral combination of Molnupiravir and Paxlovid® for the Treatment of COVID-19

Candidate-Specific Trial 9 (CST-9a): A multicentre, adaptive Phase II Platform trial to evaluate the safety, efficacy and virological response of ALG-097558 as monotherapy and in combination with Remdesivir in high-risk population for the treatment of COVID-19 disease.

Candidate-Specific Trial 9 (CST-9b): A Multicentre, Adaptive Phase II Randomised Double-Blind Placebo Controlled Trial to Evaluate the Safety, Efficacy and Virological response of ALG-097558 for the Treatment of COVID-19 disease.

ELIGIBILITY:
Master Protocol Inclusion Criteria:

1. Adults (≥18 years) with laboratory-confirmed* SARS-CoV-2 infection (PCR)
2. Ability to provide informed consent signed by study patient or legally acceptable representative
3. Women of childbearing potential (WOCBP) and male patients who are sexually active with WOCBP must agree to use a highly effective method of contraception (as outlined in the protocol) from the first administration of trial treatment, throughout trial treatment and for the duration outlined in the candidate-specific trial protocol after the last dose of trial treatment

   * If any CSTs are included in the community setting, the CST protocol will clarify whether patients with suspected SARS-CoV-2 infection are also eligible.

Standard additional criteria that may be applied per CST protocol:

Group A (severe disease) 4a. Patients with clinical status of Grades 4 (hospitalised, oxygen by mask or nasal prongs), 5 (hospitalised, on non-invasive ventilation, or high flow oxygen), 6 (hospitalised, intubation and mechanical ventilation) or 7 (ventilation and additional organ support - pressors, renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO)), as defined by the WHO clinical severity score, 9-point ordinal scale.

Group B (mild-moderate disease) 4b. Ambulant or hospitalised patients with the following characteristics peripheral capillary oxygen saturation (SpO2) >94% RA N.B. The CST protocol inclusion criteria will take precedence over the master protocol inclusion criteria.

CST-2 Inclusion Criteria:

For the purpose of the EIDD-2801 candidate-specific trial the following inclusion criteria have been amended from the Master protocol to:

1. Male or female ≥ 60 years old or ≥50 years old with at least one well controlled comorbidity: cardiovascular disease, chronic lung disease (e.g. COPD, or pulmonary hypertension), immune deficiency (taking the equivalent of 20 mg prednisone daily, chemotherapy, or immune modulating biologic therapies), diabetes (treated with insulin or oral medications), BMI≥30, or hypertension requiring medication with laboratory confirmed SARS-CoV-2 infection (PCR) .

3. Women of childbearing potential (WOCBP) and male patients who are sexually active with WOCBP must agree to use two effective methods of contraception, one of which should be highly effective (as outlined in the protocol). For women, from the first administration of trial treatment, throughout trial and up to 50 days after the last follow up visit (50 days after day 29) and for men with female partners of child bearing potential, from the first administration until 100 days after last follow up visit (100 days after day 29).

4. Group B (mild-moderate disease): Ambulant with the following characteristics peripheral capillary oxygen saturation (SpO2) >94% RA (NB this differs to the Master Protocol which also includes hospitalised patients in this group).

Additional criteria specific to this candidate are:

5. Has signs or symptoms of COVID-19 that began within 5 days of the planned first dose of study drug.

6. Is in generally good health (except for current respiratory infection) and is free of uncontrolled chronic conditions.

7. Is willing and able to comply with all study procedures and attending clinic visits through the 4th week.

8. Has someone, aged ≥ 16 living in the same household during the dosing period.

CST-6 Additional inclusion criteria:

1. Group A (severe disease). Patients with clinical status of Grades 5 (hospitalised, oxygen by mask or nasal prongs), 6 (hospitalised, on non-invasive ventilation, or high flow oxygen as defined by the WHO Clinical Progression Scale (WHO, 2020)).
2. Less than or equal to 14 days from onset of COVID-19 symptoms

CST-8 Inclusion Criteria:

1. For the purpose of CST-8, criteria 1 has been amended from the Master Protocol to:

   Adults (≥18 years) outpatients positive lateral flow test at screening or baseline Day 1, who are within 5 days of symptom onset prior to the planned first dose of study drug.
2. Criteria 3 has been amended from the Master Protocol to:

Women of childbearing potential (WOCBP) and male participants who are sexually active with WOCBP must agree to use a highly effective method of contraception (as outlined in section 5.5 of the Master Protocol) for the duration of the treatment and for six weeks following the last dose.

Additional criteria specific to CST-8 are:

* Initial onset of COVID-19 signs/symptoms within 5 days prior to the day of randomisation and at least 1 of the current specified COVID-19 signs/symptoms (listed on the NHS website) present on the day of randomisation
* Is willing and able to comply with all study procedures and attending clinic visits

CST-9a Inclusion Criteria:

For the purpose of CST-9a, criteria 1 has been amended from the Master Protocol to:

1. Adults (>/= 18 years of age) with a positive SARS-CoV-2 lateral flow test on screening or Day 1, who are at high risk (as defined in UK DHSC criteria) of progressing to severe COVID-19 disease, within 3 days of symptom onset, with at least one symptom of COVID-19 infection present on the day of randomization and are with mild- moderate disease severity at enrolment.

   Criterion 2 has been amended from the Master Protocol to:
2. Ability to provide informed consent signed by trial participant or legally acceptable representative and are willing and able to comply with all trial procedures and attending clinic visits

   Criterion 3 has been amended from the Master Protocol to:
3. Women of childbearing potential (WOCBP) and male participants who are sexually active with WOCBP must agree to use two effective methods of contraception, one of which must be highly effective for the duration of the treatment and for 90 Days following the last dose

Master Protocol Exclusion Criteria:

1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >5 times the upper limit of normal (ULN)
2. Stage 4 severe chronic kidney disease or requiring dialysis (i.e., estimated glomerular filtration rate <30 mL/min/1.73 m^2)
3. Pregnant or breast feeding
4. Anticipated transfer to another hospital which is not a study site within 72 hours
5. Allergy to any study medication
6. Patients taking other prohibited drugs (as outline in CST protocol) within 30 days or 5 times the half-life (whichever is longer) of enrolment
7. Patients participating in another CTIMP trial

N.B. The CST protocol exclusion criteria will take precedence over the master protocol exclusion criteria.

CST-9a Exclusion Criteria:

Exclusion criteria has been amended from master protocol as:

1. Prior SARS-CoV-2 infection <90 days before enrolment and/or received any COVID-19 vaccine dose <90 days before enrolment
2. Alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN) or Active Liver disease
3. History or current evidence of cirrhosis
4. Receiving dialysis or have known moderate to severe renal impairment (defined as CKD stage 4 or 5) or current acute kidney injury on most recent eGFR in the past 6 months
5. Pregnant or breast feeding
6. Anticipated transfer to another hospital which is not a trial site within 72 hours
7. Known allergy to any trial medication
8. Swallowing difficulties
9. Currently receiving ALG-097558, Paxlovid, molnupiravir or remdesivir or any SoC therapy for COVID-19 at the time of screening
10. Received sotrovimab at any point during the current SARS-CoV-2 infection
11. Oxygen saturations <94% on room air
12. Urgent or expected need for nasal high-flow oxygen therapy or positive pressure ventilation, invasive mechanical ventilation or ECMO.
13. Participants who have taken or require treatment with a comedication that is a strong CYP450 3A4 inhibitor (atazanavir, clarithromycin, itraconazole, posaconazole, voriconazole, nefazodone, nelfinavir, grapefruit juice, HIV protease inhibitors), strong CYP450 3A4 inducers (rifampin, phenytoin, carbamazepine, St. John's Wort) or sensitive substrates of CYP450 2C8 and 2B6 (repaglinide, rosiglitazone, paclitaxel, bupropion) within at least 2 weeks or 5 half-lives (whichever is longer) before the planned first dose of study drug.
14. Participating in another CTIMP trial

CST-9b Exclusion criteria:

1. Prior SARS-CoV-2 infection diagnosed <90 days before enrolment and/or received any COVID-19 vaccine dose <90 days before enrolment
2. Alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN) or Active Liver disease
3. History or current evidence of cirrhosis
4. Receiving dialysis or have known severe renal impairment defined as CKD stage 5 (an eGFR <15 mL/min/1.73 m2 at screening, or current acute kidney injury in most recent eGFR in past 6 months.
5. Pregnant or breast feeding
6. Anticipated transfer to another hospital which is not a trial site within 72 hours
7. Known allergy to any trial medication
8. Swallowing difficulties
9. Currently receiving ALG-097558, Paxlovid, molnupiravir or remdesivir or any standard of care antiviral therapy for COVID-19 at the time of screening
10. Received sotrovimab at any point during the current SARS-CoV-2 infection prior to enrolment
11. Oxygen saturations <94% on room air. NOTE: Participants on stable oxygen therapy, including use of NIPPV (non-invasive positive pressure ventilation), for a pre-existing medical condition (e.g., COPD) may be included with oxygen saturation of <94% on room air, provided there is no new increased oxygen requirement.
12. Urgent or expected need for nasal high-flow oxygen therapy or positive pressure ventilation, invasive mechanical ventilation or ECMO.
13. Participants who have taken or require treatment with a comedication that is a strong CYP450 3A4 inhibitor (atazanavir, clarithromycin, itraconazole, posaconazole, voriconazole, nefazodone, nelfinavir, grapefruit juice, HIV protease inhibitors), strong CYP450 3A4 inducers (rifampin, phenytoin, carbamazepine, St. John's Wort) or sensitive substrates of CYP450 2C8 and 2B6 (repaglinide, rosiglitazone, paclitaxel, bupropion) within at least 2 weeks or 5 half-lives (whichever is longer) before the planned first dose of study drug.
14. Participating in another CTIMP trial within 5 half-lives of the last administered dose of an investigational medicinal product.
15. Participants eligible for other antiviral treatment according to DHSC criteria, or those otherwise eligible for CST9a.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Master Protocol: Dose-finding/Phase I | 29 days from randomisation
  Determination of a dose(s) for efficacy evaluation. Dose limiting toxicities (Safety and Tolerability of drug under study - CTCAE v5 Grade ≥3 adverse events)
Master Protocol: Efficacy evaluation/Phase II - Severe patients (Group A) | 29 days from randomisation
  Determination of activity and safety.
  In severe patients (Group A): time to clinical improvement. Improvement will be determined according to the WHO Clinical Progression Scale; improvement is defined as a minimum 2-step change from randomisation in the scale up to day 29 post-randomisation.
Master Protocol: Efficacy evaluation/Phase II - Mild to moderate patients (Group B) | 15 days from randomisation
  Determination of activity and safety.
  In mild to moderate patients (Group B): pharmacodynamics of drug under study, defined as time to negative viral titres in nose and/or throat swab, measured up to 15 days post-randomisation.
CST-2 Phase I: To determine the safety and tolerability of multiple ascending doses of EIDD-2801 to recommend dose for phase II. | 7 days from randomisation
  Dose limiting toxicity (DLT) using CTCAE version 5 (grades 3 and above) over 7 days.
  CTCAE grading related to platelets and/or lymphocytes
CST-2 Phase II: To determine the ability of EIDD-2801 to reduce serious complications of COVID-19 including hospitalization, reduction in SAO2<92%, or death. | 29 days from randomisation
  Progression of disease (SpO2<92% based on at least 2 consecutive recordings on the same day) or hospitalization or death up to day 29
CST6 Phase I: To determine the safety and tolerability of multiple doses of IV Favipiravir in patients with COVID-19 | 29 days from randomisation
  Adverse events and serious adverse events
CST6 Phase I: To determine the maximum safe dose of IV Favipiravir for efficacy evaluation in phase II | 8 days from randomisation
  Dose limiting toxicities (Safety and Tolerability of IV Favipiravir- CTCAE v5 Grade ≥3 adverse events)
CST-8 Phase I: Dose Limiting Toxicities up to and including Day 11 | 11 days from randomisation
  Dose limiting toxicities (Safety and Tolerability of molnupiravir and Paxlovid® combination - CTCAE v5 Grade ≥3 adverse events) up to and including Day 11
CST-9a: Dose limiting toxicities up to and including Day 11 | 11 days from randomisation
  Dose limiting toxicities (Safety and Tolerability of ALG-097558 and ALG-097558 plus remdesivir combination - CTCAE v5 Grade ≥3 adverse events) up to and including Day 11
CST-9a: to determine the safety and tolerability of ALG-097558 and ALG-097558 plus remdesivir combination | 11 days from randomisation
  Adverse events, serious adverse events, physical findings, vital signs, ECG and laboratory parameters
CST-9a: Change in viral titre overtime following administration of ALG-097558 alone and in combination with RDV versus Standard of Care (SoC) | 11 days from randomisation
  Qualitative (and quantitative when possible) PCR for SARS-CoV-2 by nose and throat swab
CST-9a: Sustained symptom resolution | 29 days from randomisation
  Symptom resolution evaluated through questionnaires
CST-9b | 11 Days from randomisation
  AEs, SAEs
CST-9b | 11 days from randomisation
  Dose Limiting Toxicity (DLT) using CTCAE version 5 (grades 3 and above) up to and including Day 11
CST-9b | 11 days from randomisation
  Qualitative (and quantitative when possible) PCR for SARS-CoV-2 by nose and throat swab

SECONDARY OUTCOMES:
Master Protocol: Safety assessed by rate of adverse events | Up to 29 days from randomisation
  Adverse event rate according to CTCAE v5
Master Protocol: To evaluate clinical improvement | From randomisation to day 29
  Proportion of patients with clinical improvement (as defined above) at day 8, 15 and day 29.
Master Protocol: To evaluate clinical improvement using WHO clinical progression scale | From randomisation to day 15
  Change at day 8 and 15 from randomisation in the WHO Clinical Progression Scale
Master Protocol: To evaluate clinical improvement using WHO clinical progression scale | From randomisation to day 29
  Time to a one point change on the WHO Clinical Progression Scale
Master Protocol: To evaluate clinical improvement using SpO2/FiO2 | From randomisation to day 29
  The ratio of the oxygen saturation to fractional inspired oxygen concentration (SpO2/FiO2)
Master Protocol: To evaluate discharge | From randomisation to day 29
  Proportion of patient discharged at days 8, 15 and 29
Master Protocol: To evaluate admission to ICU | From randomisation to day 29
  Admission rate to ICU
Master Protocol: To evaluate safety further (WCC) | From randomisation to day 29
  White cell count on day 1, 3, 5, 8, 11 (while hospitalised); and Day 15 and 29
Master Protocol: To evaluate safety further (Hg) | From randomisation to day 29
  Haemoglobin on day 1, 3, 5, 8, 11 (while hospitalised); and Day 15 and 29
Master Protocol: To evaluate safety further (platelets) | From randomisation to day 29
  Platelets on day 1, 3, 5, 8, 11 (while hospitalised); and Day 15 and 29
Master Protocol: To evaluate safety further (creatinine) | From randomisation to day 29
  Creatinine on day 1, 3, 5, 8, 11 (while hospitalised); and Day 15 and 29
Master Protocol: To evaluate safety further (ALT) | From randomisation to day 29
  ALT on day 1, 3, 5, 8, 11 (while hospitalised); and Day 15 and 29
Master Protocol: To evaluate overall mortality | From randomisation to day 29
  Mortality at Days 8, 15 and 29. Time to death from randomisation
Master Protocol: To evaluate the number of oxygen-free days | From randomisation to day 29
  Duration (days) of oxygen use and oxygen-free days
Master Protocol: To evaluate ventilator-free days | From randomisation to day 29
  Duration (days) of mechanical ventilation and mechanical ventilation-free days
Master Protocol: To evaluate incidence of new mechanical ventilation use | From randomisation to day 29
  Incidence of new mechanical ventilation use
Master Protocol: To evaluate National Early Warning Score (NEWS)2/qSOFA | From randomisation to day 29
  NEWS2/qSOFA assessed daily while hospitalised
Master Protocol: To evaluate translational outcomes (Viral Load) | From randomisation to day 29
  Change in viral load over time
Master Protocol: To evaluate translational outcomes (Baseline SARS-COV-2) | From randomisation to day 29
  Change in viral load over time
CST-2 Additional: Pharmacokinetic Objective: To define PK of EIDD-2801 and EIDD-1931 in plasma following multiple doses administered to patients with COVID-19. | Samples collected on Day 1 and Day 5 post-randomisation
  Concentrations of EIDD-2801 and -1931 in plasma
CST-2 Additional: Virologic Objective: To assess the difference in viral clearance (time to negative PCR) between EIDD-2801 and control. | Swabs taken on Day 1 (day of randomisation), 3, 5, 8, 11, 15, 22 and 29
  Qualitative (and quantitative when possible) PCR for SARS-CoV-2 by nasal swab.
CST-2 Additional: Clinical Objective: To determine the ability of EIDD-2801 to reduce the duration of signs and symptoms of COVID-19 in patients (FLU-PRO) | From randomisation to Day 29
  Patient Reported Outcome Measures (FLU-PRO).
CST-2 Additional: Clinical Objective: To determine the ability of EIDD-2801 to reduce the duration of signs and symptoms of COVID-19 in patients (WHO Scale). | From randomisation to Day 29
  WHO Progression Scale at day 15 and 29
CST-2 Additional: Clinical Objective: To determine the ability of EIDD-2801 to reduce the duration of signs and symptoms of COVID-19 in patients (NEWS2) | From randomisation to Day 29
  NEWS2 (National Early Warning Score2) assessed during study clinic visit on days 15 and 29.
CST-2 Additional: Clinical Objective: To determine the ability of EIDD-2801 to reduce the duration of signs and symptoms of COVID-19 in patients (mortality) | From randomisation to Day 29
  Mortality at Days 15 and 29
CST-2 Additional: Clinical Objective: To determine the ability of EIDD-2801 to reduce the duration of signs and symptoms of COVID-19 in patients (death) | From randomisation to Day 29
  Time from randomisation to death
CST-6 Additional: To characterise the pharmacokinetics (PK) of multiple doses of IV Favipiravir | From randomisation to Day 8
  Plasma PK parameters of IV Favipiravir
CST-6 Additional: To investigate the ability of IV Favipiravir to reduce the duration of signs and symptoms of COVID-19 in-patients | Randomisation to Day 15 and Day 29
  WHO Progression Scale (WHO, 2020)
CST-6 Additional: To investigate the effect of IV Favipiravir on SARS-CoV-2 viral load | From randomisation to Day 29
  Viral load change from baseline over time
CST-8: Assess feasibility for late phase study by reviewing any recorded AEs and SAEs | From randomisation to Day 29
  Review of any adverse events
CST-8: Assess feasibility for late phase study by reviewing hospitalisation or death up to Day 29 | From randomisation to Day 29
  Death and hospitalisation up to Day 29
CST-8: Measure concentrations of IMP re evidence of virological efficacy | From randomisation to Day 11
  PK concentrations of both IMPs and their circulating metabolites in plasma.
CST-8: Measure PK of each drug within the combination | From randomisation to Day 11
  PK concentrations of both IMPs and their circulating metabolites in plasma.
CST8: Review evidence of virological efficacy via viral elimination slopes | From baseline to Day 11
  Qualitative (and quantitative when possible) PCR for SARS-CoV-2 by nose and throat swab
CST8: Vital signs (Heart Rate) at Screening, Baseline/Day 1, Day 3, Day 5 and Day 11 | From randomisation to Day 11
  Vital sign measure 1 heart rate (beats/min) - to be part of aggregated review of pt vitals to assess safety and tolerability.
CST-8: Vital signs (Blood Pressure) at Screening, Baseline/Day 1, Day 3, Day 5 and Day 11 | From randomisation to Day 11
  Vital sign measure 2 Blood Pressure (mmHG) - to be part of aggregated review of pt vitals to assess safety and tolerability.
CST-8: Vital signs (Respiratory Rate) at Screening, Baseline/Day 1, Day 3, Day 5 and Day 11 | From randomisation to Day 11
  Vital sign measure 3 respiratory rate (breaths/min) - to be part of aggregated review of pt vitals to assess safety and tolerability.
CST-8: Vital signs (Temperature) at Screening, Baseline/Day 1, Day 3, Day 5 and Day 11 | From randomisation to Day 11
  Vital sign measure 4 temperature (degrees c) - to be part of aggregated review of pt vitals to assess safety and tolerability.
CST-8: Vital signs (Oxygen Saturation) at Screening, Baseline/Day 1, Day 3, Day 5 and Day 11 | From randomisation to Day 11
  Vital sign measure 5 oxygen saturation (FiO2 as %) - to be part of aggregated review of pt vitals to assess safety and tolerability.
CST-9a: Measure PK of ALG-097558 plus remdesivir in plasma | Day 1 to day 3
  PK concentrations of ALG-097558 and remdesivir and metabolites in plasma
CST-9a: establish disease progression endpoints including visits to emergency department, hospitalisations, all- cause mortality | From randomisation to Day 29
  Death, hospitalisation, and hospital/GP visits
CST-9a: incidence of rebound SARS-CoV-2 infection | From randomisation to Day 29
  Proportion of participants with clinical and/or virologic rebound
CST-9a: Symptom improvement in subgroup of severely immunosuppressed participants or with high baseline viral titre | From randomisation to Day 29
  Symptom improvement evaluated through questionnaires
CST-9: Viral dynamics in subgroup of severely immunosuppressed participants or with high baseline viral titre | From randomisation to Day 29
  Viral dynamics in subgroup of severely immunosuppressed participants or with high baseline viral titre
CST-9b | 11 days from randomisation
  Plasma PK, concentrations ALG-097558 and its metabolites
CST-9b | 29 Days from randomisation
  Death, hospitalisation, and hospital/GP visits up to Day 29
CST-9b | 11 Days from randomisation
  Proportion of participants with clinical and/or virologic rebound
CST-9b | 11 Days from randomisation
  Viral dynamics in subgroup of participants with high baseline viral titre (defined as Ct value of <22)
CST-9b | 11 Days from randomisation
  Viral dynamics in subgroup of participants randomized within 3 days of symptom onset
CST-9b | 11 Days from randomisation
  Time to sustained symptom resolution (evaluated through questionnaires as a participant-reported outcome)

OTHER OUTCOMES:
CST-8: Measure PK of nirmatrelvir and ritonavir in tears, saliva and nasal secretions | From randomisation to Day 5
  Concentration of nirmatrelvir and ritonavir in non-plasma
CST-8:To characterise genetic variability in SARS-CoV-2 before and during treatment via PCR analysis | From randomisation to Day 11
  PCR analysis re Baseline and treatment emergent genetic mutations in SARS-CoV-2
CST-9a: To characterise pharmacokinetics of ALG-097558 in tears, saliva, and nasal secretions | day 1 to day 3
  Concentration of ALG-097558 in non-plasma matrices
CST-9a: To characterise genetic variability in SARS-CoV-2 before and during treatment | From randomisation to Day 11
  Baseline and treatment emergent genetic mutations in SARS-CoV-2
CST-9a: To evaluate changes in culturable virus during treatment | From randomisation to Day 11
  Viral culture from nose and throat swabs
CST-9a: To characterise time dependent changes in host response to infection or drug exposure | From randomisation to Day 11
  Translational endpoints may include transcriptomic, proteomic, genomic, and host immune response analyses, subject to the availability of qualified assays Intracellular drug metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Saye Khoo, Principal Investigator — University of Liverpool
Locations (6):
- South Africa (2):
  - Desmond Tutu Health Foundation, Cape Town
  - Ezintsha, Johannesburg
- United Kingdom (4):
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Kings College Hospital NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Master protocol publication. Data sets will be registered on the University of Liverpool Research Data Catalogue.
Supporting Information: Study Protocol
Time Frame: Master protocol published 19 June 2020
Access Criteria: Master protocol available from https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04473-1
URL: https://doi.org/10.1016/S1473-3099(22)00644-2

REFERENCES:
- [Background] Griffiths G, Fitzgerald R, Jaki T, Corkhill A, Marwood E, Reynolds H, Stanton L, Ewings S, Condie S, Wrixon E, Norton A, Radford M, Yeats S, Robertson J, Darby-Dowman R, Walker L, Khoo S; UK NIHR community. AGILE-ACCORD: A Randomized, Multicentre, Seamless, Adaptive Phase I/II Platform Study to Determine the Optimal Dose, Safety and Efficacy of Multiple Candidate Agents for the Treatment of COVID-19: A structured summary of a study protocol for a randomised platform trial. Trials. 2020 Jun 19;21(1):544. doi: 10.1186/s13063-020-04473-1. PMID 32560744
- [Background] Griffiths GO, FitzGerald R, Jaki T, Corkhill A, Reynolds H, Ewings S, Condie S, Tilt E, Johnson L, Radford M, Simpson C, Saunders G, Yeats S, Mozgunov P, Tansley-Hancock O, Martin K, Downs N, Eberhart I, Martin JWB, Goncalves C, Song A, Fletcher T, Byrne K, Lalloo DG, Owen A, Jacobs M, Walker L, Lyon R, Woods C, Gibney J, Chiong J, Chandiwana N, Jacob S, Lamorde M, Orrell C, Pirmohamed M, Khoo S; AGILE investigators. AGILE: a seamless phase I/IIa platform for the rapid evaluation of candidates for COVID-19 treatment: an update to the structured summary of a study protocol for a randomised platform trial letter. Trials. 2021 Jul 26;22(1):487. doi: 10.1186/s13063-021-05458-4. PMID 34311777
- [Result] Khoo SH, Fitzgerald R, Fletcher T, Ewings S, Jaki T, Lyon R, Downs N, Walker L, Tansley-Hancock O, Greenhalf W, Woods C, Reynolds H, Marwood E, Mozgunov P, Adams E, Bullock K, Holman W, Bula MD, Gibney JL, Saunders G, Corkhill A, Hale C, Thorne K, Chiong J, Condie S, Pertinez H, Painter W, Wrixon E, Johnson L, Yeats S, Mallard K, Radford M, Fines K, Shaw V, Owen A, Lalloo DG, Jacobs M, Griffiths G. Optimal dose and safety of molnupiravir in patients with early SARS-CoV-2: a Phase I, open-label, dose-escalating, randomized controlled study. J Antimicrob Chemother. 2021 Nov 12;76(12):3286-3295. doi: 10.1093/jac/dkab318. PMID 34450619
- [Result] Walker LE, FitzGerald R, Saunders G, Lyon R, Fisher M, Martin K, Eberhart I, Woods C, Ewings S, Hale C, Rajoli RKR, Else L, Dilly-Penchala S, Amara A, Lalloo DG, Jacobs M, Pertinez H, Hatchard P, Waugh R, Lawrence M, Johnson L, Fines K, Reynolds H, Rowland T, Crook R, Okenyi E, Byrne K, Mozgunov P, Jaki T, Khoo S, Owen A, Griffiths G, Fletcher TE; AGILE platform. An Open Label, Adaptive, Phase 1 Trial of High-Dose Oral Nitazoxanide in Healthy Volunteers: An Antiviral Candidate for SARS-CoV-2. Clin Pharmacol Ther. 2022 Mar;111(3):585-594. doi: 10.1002/cpt.2463. Epub 2021 Nov 13. PMID 34699618
- [Result] Khoo SH, FitzGerald R, Saunders G, Middleton C, Ahmad S, Edwards CJ, Hadjiyiannakis D, Walker L, Lyon R, Shaw V, Mozgunov P, Periselneris J, Woods C, Bullock K, Hale C, Reynolds H, Downs N, Ewings S, Buadi A, Cameron D, Edwards T, Knox E, Donovan-Banfield I, Greenhalf W, Chiong J, Lavelle-Langham L, Jacobs M, Northey J, Painter W, Holman W, Lalloo DG, Tetlow M, Hiscox JA, Jaki T, Fletcher T, Griffiths G; AGILE CST-2 Study Group. Molnupiravir versus placebo in unvaccinated and vaccinated patients with early SARS-CoV-2 infection in the UK (AGILE CST-2): a randomised, placebo-controlled, double-blind, phase 2 trial. Lancet Infect Dis. 2023 Feb;23(2):183-195. doi: 10.1016/S1473-3099(22)00644-2. Epub 2022 Oct 19. PMID 36272432
- [Result] FitzGerald R, Dickinson L, Else L, Fletcher T, Hale C, Amara A, Walker L, Penchala SD, Lyon R, Shaw V, Greenhalf W, Bullock K, Lavelle-Langham L, Reynolds H, Painter W, Holman W, Ewings S, Griffiths G, Khoo S. Pharmacokinetics of ss-d-N4-Hydroxycytidine, the Parent Nucleoside of Prodrug Molnupiravir, in Nonplasma Compartments of Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection. Clin Infect Dis. 2022 Aug 24;75(1):e525-e528. doi: 10.1093/cid/ciac199. PMID 35271729
- [Result] Donovan-Banfield I, Penrice-Randal R, Goldswain H, Rzeszutek AM, Pilgrim J, Bullock K, Saunders G, Northey J, Dong X, Ryan Y, Reynolds H, Tetlow M, Walker LE, FitzGerald R, Hale C, Lyon R, Woods C, Ahmad S, Hadjiyiannakis D, Periselneris J, Knox E, Middleton C, Lavelle-Langham L, Shaw V, Greenhalf W, Edwards T, Lalloo DG, Edwards CJ, Darby AC, Carroll MW, Griffiths G, Khoo SH, Hiscox JA, Fletcher T. Characterisation of SARS-CoV-2 genomic variation in response to molnupiravir treatment in the AGILE Phase IIa clinical trial. Nat Commun. 2022 Nov 26;13(1):7284. doi: 10.1038/s41467-022-34839-9. PMID 36435798
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: The AGILE Clinical Trial Platform website — http://www.agiletrial.net